CLINICAL TRIAL: NCT01909869
Title: A PILOT First-In-Man Study to Evaluate Safety and Efficacy of the EXCEL-Ⅱ With Cobalt Chromium Alloys Sirolimus Eluting Biodegradable Polymer Stent in the Treatment of Patients With de Novo Coronary Artery Lesions(CREDIT-I)
Brief Title: A Pilot First In Man Study of EXCEL-Ⅱto Treat the Patients With de Novo Coronary Artery Lesions
Acronym: CREDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2012-12
Record Dates: First submitted 2013-02-05; First posted 2013-07-29 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ischemia; Coronary Artery Disease
Keywords: MACE; TVR; MI; TLF; Death
MeSH Terms: conditions — Ischemia; Coronary Artery Disease; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EXCEL-Ⅱ (Experimental): A new Cobalt ChRomium Alloys Sirolimus Eluting BioDegradable Polymer Stent In the Treatment of Patients with de novo Coronary Artery Lesions.
  Interventions: Device: EXCEL-Ⅱ

INTERVENTIONS:
Device: EXCEL-Ⅱ — A PILOT First-In-Man Study to evaluate safety and efficacy of the EXCEL-Ⅱ with New Cobalt ChRomium Alloys Sirolimus Eluting BioDegradable Polymer Stent In the Treatment of Patients with de novo Coronary Artery Lesions
  Other Names: CREDIT-Ⅰ

SUMMARY:
One of the purpose of this study is to assess the preliminary safety and feasibility,and to provide related information and evidence for the design of the further pivotal randomized control trial.the other purpose is to assess the performace of the stent delivery system.

DETAILED DESCRIPTION:
1. Single-center, prospective, pilot study
2. De novo,coronary artery, single vessel and single lesion
3. Sample size = 45
4. Follow- up clinical or phone at 1-month,9-month and annually 2 to 5 years
5. Randomization 2:1 Angio and OCT scheduled follow-up in the hospital
6. Follow-up Angio and OCT randomized 30 patients for 4-month and 15 patiens for 12-month

ELIGIBILITY:
Inclusion Criteria:

1. 18yrs≤Age≤75yrs .
2. De novo lesion at native coronary artery.
3. Single target vessel and single target lesion.
4. Lesion length ≤32mm.
5. RVD 2.5mm～4.0mm.
6. DS%≥70% by visual estimation.
7. Target lesion could be covered by only one stent.
8. Subjects are willing to follow the specified requirements follow-up.
9. A process by which a subject voluntarily confirms his or her willingness to participate in a particular trial, after having been informed of all aspects of the trial that are relevant to the subject's decision to participate. Informed consent is documented by means of a written, signed and dated informed consent form.

Exclusion Criteria:

1. AMI within one week.
2. CTO(TIMI0),LM lesion,ostial lesion,graft vessel lesion,bifurcation (side branch RVD≥2.5mm),ISR,mutivessel disease need to be treated.
3. Severe calcified lesion unable to predilate.
4. extremely tortuous proximal to the lesion that is inadequate to stent delivery.
5. NYHA≥Ⅲ or LVEF≤40%.
6. Prior stenting within 1 year.
7. Pregnancy or lactation, and plan in postoperative pregnancy or lactation.
8. Subjects had bleeding tendency or blood coagulation dysfunction or PCI contraindications, or anticoagulant therapy taboo or can't continue DAPT healers at least 1 year.
9. There are other diseases (such as cancer,malignant tumor ,congestive heart failure,organ transplantation or candidate) or abuse history (alcohol cocaine heroin, etc.), scheme compliance is poor, interference related data explanation or the limited life (< 1 year).
10. To aspirin heparin clopidogrel cobalt chromium alloy rapamycin PLA polymer contrast agent of one of allergy.
11. Serious liver and kidney function is not complete person.
12. The investigators think that do not fit to enroll the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint(MACE) | 30days(MACE)
  Device oriented cardiovascular endpoint at 30-day (MACE) defined as the composite of Cardiac Death,Myocardial Infarction(Q and non-Q) or Ischemia-driven Target Lesion Revascularization

SECONDARY OUTCOMES:
Secondary endpoint | 5 years (Follow-up)
  In-stent Late Lumen Loss at 4-month and 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Han y ling, PhD, Principal Investigator — Shenyang Northern Hospital
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China